CLINICAL TRIAL: NCT03769506
Title: A Phase 3, Randomized, Double-Arm, Open-Label, Controlled Trial of ASP-1929 Photoimmunotherapy Versus Physician's Choice Standard of Care for the Treatment of Locoregional, Recurrent Head and Neck Squamous Cell Carcinoma in Patients Who Have Failed or Progressed On or After at Least Two Lines of Therapy, of Which at Least One Line Must Be Systemic Therapy
Brief Title: ASP-1929 Photoimmunotherapy (PIT) Study in Recurrent Head/Neck Cancer for Patients Who Have Failed at Least Two Lines of Therapy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rakuten Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASP-1929-301
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
Keywords: Rakuten Medical; ASP-1929; PIT; Photoimmunotherapy; HNC; HNSCC; Head and neck; EGFR; Cetuximab; Erbitux; RM-1929
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- ASP-1929 Photoimmunotherapy (Experimental): Use of ASP-1929 Photoimmunotherapy
  Interventions: Combination Product: ASP-1929 Photoimmunotherapy
- Physician's Choice SOC (Active Comparator): docetaxel, cetuximab, methotrexate, paclitaxel
  Interventions: Drug: Physician's Choice SOC

INTERVENTIONS:
Combination Product: ASP-1929 Photoimmunotherapy — Use of ASP-1929 PIT therapy
  Arms: ASP-1929 Photoimmunotherapy
Drug: Physician's Choice SOC — docetaxel, cetuximab, methotrexate, paclitaxel
  Arms: Physician's Choice SOC

SUMMARY:
A Phase 3, Randomized, Double-Arm, Open-Label, Controlled Trial of ASP-1929 vs Physician's Choice Standard of Care for the Treatment of Locoregional, Recurrent Head and Neck Squamous Cell Carcinoma in Patients Who Have Failed or Progressed On or After at Least Two Lines of Therapy

DETAILED DESCRIPTION:
The study will have an Experimental Arm and a Control Arm.

Experimental Arm:

Patients may receive repeated ASP-1929 PIT interventions for up to a maximum of 8 cycles within a period of up to 12 months after randomization until the patient has complete remission, progressive disease that is no longer amendable to study treatment, patient experiences intolerable side effects, patient discontinues study treatment, or chooses to withdraw. Repeat ASP-1929 treatment cycles will be administered no less than 4 weeks from the previous ASP-1929 infusion.

Control Arm:

Patients may be treated with physician's choice standard of care until the patient has progressive disease, patient experiences intolerable side effects, discontinues study treatment, or chooses to withdraw.

ELIGIBILITY:
Overall Inclusion Criteria:

* Have a histologically confirmed locoregional persistent, recurrent or second primary squamous cell carcinoma of the head and neck, not amenable to curative treatment
* Have failed or progressed on or after at least 2 lines of therapy for squamous cell carcinoma of the head and neck, one of which must be prior systemic platinum-based chemotherapy
* Have completed prior curative radiation therapy for treatment of their head and neck region
* Have locoregional head and neck tumor site(s) that are all accessible to light illumination
* Have target tumors that are clearly measurable by contrast enhanced CT scan, or MRI scan with gadolinium if CT scan is not adequate or the patient has an allergy to CT contrast media.
* Have a life expectancy of > 6 months, based on Investigator judgment
* Male participants must agree to use contraception during the treatment period and for at least 6 months after the last ASP-1929 infusion
* Female patients of childbearing potential must not be pregnant or breastfeeding and agree to follow the contraceptive guidance during the treatment period and for at least 6 months after the last dose of trial intervention and must refrain from breastfeeding for at least 2 months after the last ASP-1929 infusion
* Have an Eastern Cooperative Oncology Group (ECOG) score of 0 or 1

Overall Exclusion Criteria:

* Have a history of significant (>= Grade 3) cetuximab infusion reactions
* Have been treated with prior systematic chemotherapy or targeted small molecule therapy or radiation therapy within 2 weeks of trial Day 1 or not recovered from adverse events due to a previously administered agent
* Have been treated with an anticancer monoclonal antibody therapy within 4 weeks of trial Day 1 or have not recovered from adverse events due to previously administered agent
* Have been treated with an investigational agent or intervention within 4 weeks of trial Day 1 or have not recovered from adverse events, due to previously administered agent or intervention
* Have a present history of distant metastatic disease (M1)
* Have an active undergoing treatment or have a diagnosis of an active cancer other than nonmelanoma skin cancer or HNSCC
* Have a tumor in enhanced CT or MRI scan invading a major blood vessel, unless the vessel has been embolized, stented or surgically ligated to prevent potential bleeding from a blood vessel
* Have impaired hepatic function
* Have impaired renal function
* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with trial requirements
* Have been previously treated or randomized to any trial using ASP-1929 or RM-1929 PIT as the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  PFS, defined as the time from randomization to the first occurrence of disease progression (PD), as determined by the Central Radiographic Review according to RECIST 1.1 with modifications, or death from any cause, whichever occurs first.
Overall Survival (OS) | 24 months
  OS, defined by the time interval between the patient randomization and death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 24 months
  ORR, defined by the percentage of patients with the best overall response of complete response (CR) or partial response (PR) by RECIST 1.1 with modifications.
Duration of Response (DoR) | 24 months
  DoR, defined as the time from first objective response (CR or PR) to the date of the first documented tumor progression, as determined by Central Radiographic Review according to RECIST 1.1 criteria with modifications or date of death due to any cause, whichever occurs first.
Event-Free Survival (EFS) | 24 months
  EFS, defined as the time interval from randomization to a >20% increase in tumor size from baseline (CT or MRI scan at screening) by Central Radiographic Review according to RECIST 1.1 with modifications, development of new locoregional disease, distant metastatic disease, or death, whichever occurs first.
Eastern Cooperative Oncology Group (ECOG) performance status | 24 months
Quality of Life (QoL) assessment - EORTC QLQ-C30 | 24 months
  Change from baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30). EORTC QLQ-C30 is a 30-item questionnaire developed to assess QoL of head and neck cancer participants and consists of five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health status scale, and a number of single items assessing additional symptoms commonly reported by cancer patients (dyspnoea, loss of appetite, insomnia, constipation and diarrhea) and perceived financial impact of the disease. It has four-point scales for the first 28 items. The minimum value is 1 and maximum value is 4. Higher scores mean a worse outcome. Overall health was evaluated as a 7-point response scale as the other two questions in that scale. The minimum value is 1 and maximum value is 7. Higher scores mean a better outcome.
Quality of Life (QoL) assessment - EORTC QLQ H&N 35 | 24 months
  Change from baseline in EORTC head and neck specific module (EORTC QLQ H&N 35). EORTC QLQ-H&N35 is a 35-item questionnaire developed to assess QoL of head and neck cancer participants and consists of 7 multiple-item scales that assess the symptom of pain, swallowing, senses (taste/smell), speech, social eating, social contact and sexuality. Also, six single-item scales are included to survey the presence of symptomatic problems associated with teeth, mouth=opening, dry mouth, sticky saliva, coughing, and feeling ill. The minimum value is 1 and maximum value is 4. It has 2-point scales for the last 5 items. The minimum value is 1 and maximum value is 2. For all items and scales, high scores indicate more problems.
Quality of Life (QoL) assessment - EQ 5D-5L | 24 months
  Change from baseline in EuroQol 5-Dimension 5-Level (EQ 5D-5L) Questionnaire. EQ-5D-5L is a 5-dimension (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) questionnaire developed to assess the patient-generated health state index score from the societal perspective and subjective perceived health. For each dimension, levels of perceived problems are coded from level 1 (minimum) to level 5 (maximum): no problems (1), slight problems (2), moderate problems (3), severe problems (4), and extreme problems/inability (5). A second part of the questionnaire provides a visual analogue scale (VAS) for individually perceived health from 0 to 100 (corresponding to the worst to the best imaginable health).
Population Pharmacokinetics (PK) of ASP-1929 | 12 months
  Estimate covariate effects of ASP-1929 PK through compartmental PK modeling.
Presence of Anti-Drug Antibodies (ADA) of ASP-1929 | 24 months
Complete Response (CR) | 24 months
  CR, defined as the proportion of patients with tumor response of CR, as determined by Central Radiographic Review according to RECIST 1.1 with modifications.
Complete Response by Biopsy (CRb) | 24 months
  CR by histopathologic biopsy of target tumor(s) and a repeated confirmatory histopathologic CR biopsy at least 3 months after initial CR histopathologic biopsy of the target tumor(s) for patients who demonstrate a clinical CR but not an image CR per RECIST 1.1 with modifications, as determined by the Investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Chen, MD, Study Director — Rakuten Medical
Locations (21):
- United States (7):
  - Cancer Clinic, Miami, Florida
  - Cancer Clinic, Tampa, Florida
  - Cancer Clinic, Atlanta, Georgia
  - Cancer Clinic, Lexington, Kentucky
  - Cancer Clinic 1, Philadelphia, Pennsylvania
  - Cancer Clinic 2, Philadelphia, Pennsylvania
  - Cancer Clinic, Houston, Texas
- India (7):
  - Cancer Clinic, Vadodara, Gujarat
  - Cancer Clinic, Bangalore, Kamataka
  - Cancer Clinic, Kochi, Kerala
  - Cancer Clinic, Chennai, Tamil Nadu
  - Cancer Clinic, Hyderabad, Telangana
  - Cancer Clinic, Kolkata, West Bengal
  - Cancer Clinic, Mumbai
- Japan (4):
  - Cancer Clinic, Nagoya, Aichi-ken
  - Cancer Clinic, Sapporo, Hokkaido
  - Cancer Clinic, Okayama, Okayama-ken
  - Cancer Clinic, Chuo-ku, Tokyo
- Taiwan (3):
  - Cancer Clinic, Taichung
  - Cancer Clinic, Taipei
  - Cancer Clinic, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kobayashi H, Furusawa A, Rosenberg A, Choyke PL. Near-infrared photoimmunotherapy of cancer: a new approach that kills cancer cells and enhances anti-cancer host immunity. Int Immunol. 2021 Jan 1;33(1):7-15. doi: 10.1093/intimm/dxaa037. PMID 32496557
- [Background] Kobayashi H, Choyke PL. Near-Infrared Photoimmunotherapy of Cancer. Acc Chem Res. 2019 Aug 20;52(8):2332-2339. doi: 10.1021/acs.accounts.9b00273. Epub 2019 Jul 23. PMID 31335117
- [Derived] Magagoum SH, Biteghe FAN, Siwe GT, Lang D, Lekena N, Barth S. SNAP-Tag-Based Recombinant Photoimmunotherapeutic Agents for the Selective Detection and Killing of Light-Accessible Melanotransferrin-Expressing Melanoma and Triple-Negative Breast Cancer. Cancer Med. 2025 May;14(9):e70912. doi: 10.1002/cam4.70912. PMID 40326388